CLINICAL TRIAL: NCT05630729
Title: Living With CKD: An E-Learning Platform for Adolescents With CKD About the Disease and Its Management
Acronym: CKD Delp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R44DK108421 (NIH)
Record Dates: First submitted 2020-06-15; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Chronic Kidney Diseases; Chronic Kidney Disease stage3; Chronic Kidney Disease stage4; Chronic Kidney Disease Stage V; Chronic Kidney Disease Stage 5; Chronic Kidney Disease Stage 2; Chronic Kidney Disease, Stage I; Chronic Kidney Disease, Stage IV (Severe); Pediatric Kidney Disease
Keywords: Chronic Kidney Disease; Disease Self-Management; Adolescent Health
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My Kidney Guru Intervention (Other): Youth Participants with CKD will complete the 9 My Kidney Guru modules over the 6-month intervention period, at a rate of approximately one module every 2-3 weeks. Parent participants will complete the parent module within the first t2 weeks of the intervention period, and to review the remaining youth modules by the end of the trial period. Participants will complete outcomes measures within 1 month prior to beginning the intervention. Software usage data will be gathered regarding fidelity and dosage of the My Kidney Guru intervention. Within 1 month of completing the intervention period, participants will complete the same set of outcomes assessments, along with an evaluation survey of the intervention. Once post-intervention data collection has been completed and the intervention period has ended, participants will participate in a 45 minute follow up Web-Ex focus group to provide feedback on their experiences with My Kidney Guru and collect additional suggestions for improvement.
  Interventions: Other: My Kidney Guru

INTERVENTIONS:
Other: My Kidney Guru — My Kidney Guru is a program that will offer pediatric patients with CKD developmentally appropriate, interactive, and engaging instruction and practice opportunities to build knowledge and skills to manage CKD.

SUMMARY:
Leveraging a unique combination of synchronized web and mobile applications, this 3 year SBIR Phase II project will fully develop and pilot test My Kidney Guru-a program that will offer pediatric patients with CKD developmentally appropriate, interactive, and engaging instruction and practice opportunities to build knowledge and skills to manage CKD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a progressive condition, characterized by an irreversible deterioration of renal function that gradually progresses to end-stage renal disease, requiring dialysis or kidney transplant. CKD and its co-morbidities (e.g., hypertension, anemia, acidosis, and metabolic bone disease) require strict treatment adherence to halt progression and improve outcomes. Unfortunately, the majority of pediatric patients with CKD do not adhere to their medical regimen. This non-adherence can have devastating consequences such as renal failure, kidney transplant rejection, and even death. Research underscores how a lack of information or misinformation undermines adherence, and how static educational materials are not sufficient to ensure adherence to treatment. In order to optimize adherence, there is a need for educational programs to include a behavioral self-management component. Moreover, web-based tools are well accepted among CKD patients and online education has been shown to significantly improve health outcomes for adults with chronic illness. Leveraging a unique combination of synchronized web and mobile applications, this 3 year SBIR Phase II project will fully develop and pilot test My Kidney Guru-a program that will offer pediatric patients with CKD developmentally appropriate, interactive, and engaging instruction and practice opportunities to build knowledge and skills to manage CKD. The contextually-relevant program will include personalized tools for self-monitoring and self-management including coping strategies for managing psychological and psychosocial aspects of a chronic condition. The proposed project will accomplish three specific aims: (1) Fully develop the program, including nine modules, using an iterative user-centered development-testing-revision process to ensure the software achieves optimal usability for intended end users. (2) Conduct a pilot efficacy study to assess the program's impact for improving adolescents' CKD and self-management knowledge, treatment adherence, transition readiness, self-management skills, self-efficacy, and quality of life. Adolescents with CKD will complete the nine modules over a 6-month intervention period. Parents of adolescents will review the parent module at the beginning of the trial and the youth modules at the end of the trial. Investigators expect adolescents to report significant improvements in all areas. Lastly, investigators will (3) prepare the product for commercialization by conducting focus groups with healthcare providers to review the program and gather feedback regarding implementation in healthcare delivery settings. In preparation for Phase III commercial launch, investigators will finalize revisions and reporting functions, and integrate e-commerce functions into the website. The proposed My Kidney Guru program will directly address the need for innovative solutions to effectively increase treatment adherence using a dynamic education and self-management program designed specifically to meet the needs of adolescents with CKD. Greater adherence and self-management skill will translate into significant benefits in the well-being of these youth, including lower risk for medical complications and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 13-25 years old
* Been in Stage 1-5 CKD for at least 3 months or <1 year post transplant
* English Language fluency
* No significant intellectual or developmental delays

Exclusion Criteria:

* Adolescents who participated in the Phase I feasibility testing or Phase II usability testing will be excluded from the pilot test due to their familiarity with the proposed product.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Self-Management and Transition to Adulthood Treatment Questionnaire at 6 months | 6 months apart, as pre- and post-tests
  Both parents and adolescents will complete this 18-item measure, rating the extent to which youth are ready to transition to self-care and manage their health-related needs independently. Items assess adolescents' independence in scheduling doctor's appointments, remembering to take medication, finding answers to health-related questions, knowledge of their condition, and how easy/difficult these tasks are for the youth. Responses range from 0 (Never, Very Hard, or Nothing) to 5 (Always, Very Easy, or A Lot). Total scores range from 0 to 90. Higher scores reflect better outcomes.

SECONDARY OUTCOMES:
Change from Baseline Beliefs about Dietary Compliance scale at 6 months | 6 months apart, as pre- and post-tests
  This modified measure contains 9 items, on which adolescents and their parents report on their perceptions of the benefits and barriers of adherence to the condition treatment regimen. Responses range from 0 (strongly disagree) to 4 (strongly agree). Total scores range from 0 to 36. Higher scores reflect greater perceived benefits.
Change from Baseline Chronic Kidney Disease Self-Efficacy Instrument at 6 months | 6 months apart, as pre- and post-tests
  Adolescents will complete this 25-item reporting their self-confidence in managing their condition, including self-confidence in (a) managing the disease autonomously, (b) integrating treatment requirements to fit new situations or social activities, (c) finding solutions to CKD-related problems, and (d) finding social support when needing help. Responses range from 1 (not at all confident) to 10 (totally confident). Total scores range from 25 to 250. Higher scores reflect improved outcomes.
Change from Baseline Self-Efficacy for Managing Chronic Disease Scale at 6 months | 6 months apart, as pre- and post-tests
  Adolescents will report on condition self-management by responding to 6 items reporting their confidence and ability to observe and understand symptoms. Responses range from 0 (not at all confident) to 10 (totally confident). Total scores range from 0 to 60. Higher scores reflect improved outcomes.
Change from Baseline Illness Perception Questionnaire-Revised at 6 months | 6 months apart, as pre- and post-tests
  Adolescent participants report their perceptions of the severity of their condition. These items assess the extent to which a patient believes their condition to be serious and to have major consequences on his/her life. Responses range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 6 to 30. Higher scores reflect worse outcomes.
Change from Baseline Center for Epidemiologic Studies Depression Scale at 6 months | 6 months apart, as pre- and post-tests
  Adolescent participants respond to the this 20-item measure rating how often they experienced symptoms associated with depression over the past week, including poor sleep, loss of appetite, and loneliness. Responses range from 1 (rarely) to 4 (all of the time). Total scores range from 20 to 80. Higher scores reflect worse outcomes.
Change from Baseline Kidney Disease and Quality of Life-Short Form at 6 months | 6 months apart, as pre- and post-tests
  Adolescent participants will complete a subset of 19 items modified to be more general and applicable to any medical condition. These items comprise subscales that assess patients' symptoms, burden of condition in interfering with life, cognitive functioning, social support, and difficulty sleeping. Items are scored based on the configuration of the item (e.g., frequency of behavior, 1-non to 6-very severe). Total scores range from 15-91. Higher scores indicate worse outcomes.
Change from Baseline Knowledge of My Kidney Guru at 6 months | 6 months apart, as pre- and post-tests
  On this measure, both parent and adolescent participants complete a 30 item multiple choice questionnaire designed to assess their knowledge of information learned in the My Kidney Guru program. Each item is worth 0 to 1 point. Total scores range from 0 to 20. Higher scores reflect better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Childress, PHD, Principal Investigator — 3- C Institute for Social Development, dba 3C Institute; Maria Ferris, MD, PHD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - 3C Institute, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No